CLINICAL TRIAL: NCT00455975
Title: Phase II Trial of High-Dose Bevacizumab in the Treatment of Patients With Advanced Clear Cell Renal Carcinoma
Brief Title: High-dose Bevacizumab in Advanced Renal Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 43; AVF 3913s
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Renal Cancer; Kidney Cancer
Keywords: Kidney Cancer; Renal Cancer; Clear Cell Carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Adenocarcinoma, Clear Cell | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly Avastin (Experimental): Bevacizumab 15mg/kg IV weekly until progressive disease or toxicity
  Interventions: Drug: Bevacizumab
- Bi-weekly Avastin (Experimental): Bevacizumab 15mg/kg IV every 2 weeks until progressive disease or toxicity
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin

SUMMARY:
This trial will examine the effectiveness and the side effects of 2 higher dosing schedules of bevacizumab in patients that have advanced clear cell renal carcinoma.

DETAILED DESCRIPTION:
Bevacizumab is considered a targeted drug. Targeted drugs act on specific receptors on a cell. Bevacizumab blocks receptors that help cancer cells develop blood supplies so that the cancer can grow. These specific receptors are found in greater numbers in kidney cancer. In that regard bevacizumab will be tested in 2 doses that are higher than non-kidney cancer treatments with bevacizumab.

One group of patients will receive bevacizumab at 15 mg per kg by vein every 2 weeks. A total of 75 patients will be treated with this dose.

If this dose is well tolerated a second group of patients will receive bevacizumab at 15mg per kg by vein weekly.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic or unresectable locally recurrent clear cell renal carcinoma
* Previous kidney removal is required except if the primary tumor was smaller than 5 cm or there was extensive liver or bone metastasis
* Patients may have received a maximum of 1 prior systemic treatment of immunotherapy (Interferon, IL-2), chemotherapy, or combination chemo+immunotherapy for metastatic disease.
* No prior bevacizumab
* Measurable disease
* Adequate liver and kidney function
* Age 18 and older

Exclusion Criteria:

* Acute MI within the past 6 months
* Uncontrolled high blood pressure or history of hypertensive crisis
* Clinically significant cardiovascular disease
* Active brain cancer
* Meningeal metastasis
* Pregnant or lactating women
* Prior treatment for another cancer less than 5 years ago
* No diseases of the central nervous system (eg. uncontrolled seizures, strokes or TIAs
* No bleeding from the mouth, rectum or coughing up blood or history of other bleeding or clotting disorders
* No history of deep vein thrombosis less than 12 months ago or are currently requiring full dose anticoagulation
* No major surgical procedures, open biopsies or traumatic injury in past 28 days
* No patients with peg tubes or feeding tubes
* No patients with non healing wounds, ulcers or long bone fractures
* No history of abdominal fistulas, gastrointestinal perforation or intrabdominal abscess within 6 months
* No symptomatic peripheral vascular disease

Please note: there are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Methodist Cancer Center, Omaha, Nebraska
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Started | 58 | 61
Completed | 40 | 40
Not Completed | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Avastin | Bi-weekly Avastin | Total
Number analyzed (Participants) | 58 | 61 | 119
Age, Continuous [Median (Full Range); unit: years] | 65 [44 to 88] | 60 [40 to 88] | 63 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 34 | 44 | 78
Region of Enrollment [Number; unit: participants]
  United States | 58 | 61 | 119

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival is measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death on study. Progression is defined in RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 18 months (expected)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Number analyzed (Participants) | 58 | 61
months | 6.0 [3.5 to 9.1] | 5.7 [3.6 to 9.2]

2. Secondary Outcome: Overall Survival (OS)
Description: Measured from date of study entry to date of death due to any cause.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Number analyzed (Participants) | 58 | 61
months | 26.9 [12.9 to NA] — Upper bound of 95% confidence interval not reached at this time point | 18.4 [12.0 to 28.9]

3. Secondary Outcome: Objective Response Rate
Description: The number of patients with observed complete response [CR] or partial response [PR]. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Number analyzed (Participants) | 58 | 61
participants | 9 | 6

4. Secondary Outcome: Overall Tolerability and Toxicity of High-dose Bevacizumab
Description: Number of patients treated with high-dose bevacizumab experiencing Grade 3/4, treatment-related toxicities
Time Frame: 18 months
Population: All patients treated with Bevacizumab therapy were assessed for Grade 3/4 toxicities
Measure: Number; unit: participants
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Number analyzed (Participants) | 58 | 61
participants
  Anemia | 2 | 5
  Thrombocytopenia | 1 | 0
  Hypertension | 13 | 14
  Proteinuria | 17 | 12
  Dyspnea | 4 | 3
  Fatigue | 0 | 4
  Nausea/vomiting | 0 | 4
  Anorexia | 1 | 2
  Headache | 1 | 1
  Confusion | 0 | 2
  Allergic/hypersensitivity reaction | 1 | 1
  Hemorrhage | 3 | 1
  Thrombosis/embolism | 1 | 3
  Arthralgia | 1 | 1
  Neuropathy/sensory | 1 | 0
  Colitis | 1 | 0
  Gastroenteritis | 0 | 1
  Renal failure | 0 | 1
  Myocardial infarction | 1 | 0
  Stroke | 1 | 0
  Tracheoesophageal fistula | 1 | 0

ADVERSE EVENTS:
Arm/Group | Weekly Avastin | Bi-weekly Avastin
Serious Adverse Events (participants affected / at risk) | 33/58 | 35/61
Other Adverse Events (participants affected / at risk) | 58/58 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weekly Avastin (N=58) | Bi-weekly Avastin (N=61)
Dehydration (Metabolism and nutrition disorders) | 2 | 2
General disorders and administration site conditions - Other, disease progression (General disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 2 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 0 | 2
Stroke (Nervous system disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Bone infection (Infections and infestations) | 0 | 1
Cardiac disorders - Other, ischemia (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Esophageal fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1 | 0
Heart Failure (Cardiac disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other, gastroenteritis (Infections and infestations) | 0 | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 0 | 1
Musculoskeletal and connective tissue disorders - Other, lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other, renal failure (Renal and urinary disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, chronic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weekly Avastin (N=58) | Bi-weekly Avastin (N=61)
FATIGUE (General disorders) | 37 | 50
PROTEINURIA (Renal and urinary disorders) | 34 | 39
NAUSEA (Gastrointestinal disorders) | 21 | 22
Anorexia (Metabolism and nutrition disorders) | 14 | 24
HEADACHE (Nervous system disorders) | 18 | 17
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 19
HYPERTENSION (Vascular disorders) | 30 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 21
Constipation (Gastrointestinal disorders) | 10 | 16
VOMITING (Gastrointestinal disorders) | 8 | 15
Abdominal pain (Gastrointestinal disorders) | 7 | 15
Rash (Skin and subcutaneous tissue disorders) | 8 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 11
Diarrhea (Gastrointestinal disorders) | 0 | 16
Fever (General disorders) | 5 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 15
Edema limbs (General disorders) | 0 | 13
Allergic reaction (Immune system disorders) | 4 | 9
Insomnia (Psychiatric disorders) | 4 | 9
Dizziness (Nervous system disorders) | 0 | 12
hyperkalemia (Metabolism and nutrition disorders) | 0 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 5
Oral pain (Gastrointestinal disorders) | 4 | 6
Chills (General disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Creatinine increased (Investigations) | 0 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 6
Edema (General disorders) | 4 | 5
Depression (Psychiatric disorders) | 3 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 8
Renal and urinary disorders - Other, urinary hemorrhage (Renal and urinary disorders) | 3 | 5
Non-cardiac chest pain (General disorders) | 1 | 7
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Respiratory, thoracic and mediastinal disorders - Other, sinus drainage (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Alkaline phosphatase increased (Investigations) | 0 | 6
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 0
Mucositis (Gastrointestinal disorders) | 0 | 5
Weight loss (Investigations) | 0 | 5
Rhinitis infective (Infections and infestations) | 2 | 3
Tremor (Nervous system disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.